CLINICAL TRIAL: NCT02484066
Title: Diagnostic Value of Virtual Bronchoscopic Navigation (VBN) Combined With Endobronchial Ultrasound (EBUS) With a Guide Sheath (GS) for Peripheral Pulmonary Lesions (PPLs) Without Fluoroscopy: a Randomized Controlled Trial
Brief Title: VBN-EBUS-GS-TBLB With or Without Fluoroscopy for the Diagnosis of PPLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiayuan Sun (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director, Department of Endoscopy, Shanghai Chest Hospital, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE201503
Record Dates: First submitted 2015-06-16; First posted 2015-06-29 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Lung Cancer
Keywords: Virtual bronchoscopic navigation; Endobronchial ultrasound; Guide Sheath; Transbronchial biopsy; Peripheral pulmonary lesions
MeSH Terms: conditions — Lung Neoplasms | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VBN-EBUS-GS group (Experimental): Fluoroscopy are not used in this group. EBUS and GS are inserted into bronchi in the assistance of VBN. The EBUS probe and GS are confirmed to reach the lesion by EBUS images alone, cytologic and pathologic specimens are obtained without fluoroscopic guidance.
  Interventions: Device: VBN; Device: EBUS-GS
- VBN-EBUS-GS-X-ray group (Active Comparator): EBUS and GS are inserted into bronchi in the assistance of VBN. The EBUS probe and GS are confirmed to reach the lesion by EBUS images and radiograph fluoroscopy, cytologic and pathologic specimens are obtained with fluoroscopic guidance.
  Interventions: Device: VBN; Device: EBUS-GS; Device: X-ray

INTERVENTIONS:
Device: VBN — VBN is carried out by a VBN software（DirectPath; Olympus, Japan) which can automatically create virtual bronchoscopic images.
Device: EBUS-GS — EBUS is performed using an endoscope ultrasound system , which is equipped with a 20-MHz mechanical radial-type probe (UM-S20-17S;Olympus) with an external diameter of 1.4 mm and a GS (K-201; Olympus).
Device: X-ray — The radiograph fluoroscopy are performed when the probe and GS are confirmed to reach the lesion by EBUS images ,cytologic and pathologic specimens are obtained under fluoroscopic guidance.
  Arms: VBN-EBUS-GS-X-ray group

SUMMARY:
The purpose of this study is to evaluate the feasibility, efficacy and safety of transbronchial lung biopsy (TBLB) and bronchial brushing by using virtual bronchoscopic navigation (VBN) combined with endobronchial ultrasound (EBUS) and a Guide Sheath (GS) for the diagnosis of peripheral pulmonary lesions (PPLs) without radiographic fluoroscopy.

DETAILED DESCRIPTION:
The investigators evaluate the feasibility, efficacy and safety of transbronchial lung biopsy (TBLB) and bronchial brushing by using virtual bronchoscopic navigation (VBN) combined with endobronchial ultrasound (EBUS) and a Guide Sheath (GS) as a guide for diagnosing peripheral pulmonary lesions (PPLs) without radiographic fluoroscopy.The study is designed as a three centers prospective randomized controlled trial.The participating centers are Department of endoscopy , Shanghai chest Hospital, Shanghai JiaoTong University, China. Department of endoscopy, National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, China. Department of Respiratory Medicine, The First Affiliated Hospital of Guangzhou Medical University, China. Patients are divided into two groups, VBN-EBUS-GS-X-ray group and VBN-EBUS-GS group. Each subject will be randomized to each group. The study is expected to enroll 436 patients at 3 centers.

ELIGIBILITY:
Inclusion Criteria:

* Individuals eligible for inclusion are patients that the CT scan appearance of the PPLs showed the longest diameter was more than 8mm and non GGO lesions.

Exclusion Criteria:

1. Absence of bronchus leading to or adjacent to the lesion from CT scan
2. Refusal of participation
3. Severe cardiopulmonary dysfunction and other indications that can't receive bronchoscopy
4. Presence of concomitant endobronchial lesion during the brochoscopy procerdure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
The difference of diagnostic value of VBN-EBUS-GS-TBLB with fluoroscopy as compared to VBN-EBUS-GS-TBLB | one year
  The diagnostic value means sensitivity and specificity in two groups

SECONDARY OUTCOMES:
The difference of operation time of VBN-EBUS-GS-TBLB with fluoroscopy as compared to VBN-EBUS-GS-TBLB | one year
  The operation time includes total operation time,total GS time and total EBUS time
The difference of complications of VBN-EBUS-GS-TBLB with fluoroscopy as compared to VBN-EBUS-GS-TBLB | one year
  Complications mean a composite of operation-related serious adverse events (pneumothorax, bleeding, etc.) during and after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Sun Jiayuan, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

REFERENCES:
- [Background] Kurimoto N, Miyazawa T, Okimasa S, Maeda A, Oiwa H, Miyazu Y, Murayama M. Endobronchial ultrasonography using a guide sheath increases the ability to diagnose peripheral pulmonary lesions endoscopically. Chest. 2004 Sep;126(3):959-65. doi: 10.1378/chest.126.3.959. PMID 15364779
- [Background] Yoshikawa M, Sukoh N, Yamazaki K, Kanazawa K, Fukumoto S, Harada M, Kikuchi E, Munakata M, Nishimura M, Isobe H. Diagnostic value of endobronchial ultrasonography with a guide sheath for peripheral pulmonary lesions without X-ray fluoroscopy. Chest. 2007 Jun;131(6):1788-93. doi: 10.1378/chest.06-2506. PMID 17565021
- [Background] Yamada N, Yamazaki K, Kurimoto N, Asahina H, Kikuchi E, Shinagawa N, Oizumi S, Nishimura M. Factors related to diagnostic yield of transbronchial biopsy using endobronchial ultrasonography with a guide sheath in small peripheral pulmonary lesions. Chest. 2007 Aug;132(2):603-8. doi: 10.1378/chest.07-0637. Epub 2007 Jun 15. PMID 17573504
- [Background] Steinfort DP, Khor YH, Manser RL, Irving LB. Radial probe endobronchial ultrasound for the diagnosis of peripheral lung cancer: systematic review and meta-analysis. Eur Respir J. 2011 Apr;37(4):902-10. doi: 10.1183/09031936.00075310. Epub 2010 Aug 6. PMID 20693253
- [Background] Ishida T, Asano F, Yamazaki K, Shinagawa N, Oizumi S, Moriya H, Munakata M, Nishimura M; Virtual Navigation in Japan Trial Group. Virtual bronchoscopic navigation combined with endobronchial ultrasound to diagnose small peripheral pulmonary lesions: a randomised trial. Thorax. 2011 Dec;66(12):1072-7. doi: 10.1136/thx.2010.145490. Epub 2011 Jul 11. PMID 21749984